CLINICAL TRIAL: NCT05702060
Title: Comparison of raDiatiOn Exposure to Operators in Coronary Angiography and Percutaneous Coronary Intervention Between Right Conventional and Left Distal Radial artEry Approach: Multicenter, Randomized Study
Brief Title: Randomized Comparison of Radiation Exposure to Operators in Coronary Intervention Between Right Radial and Left DRA
Acronym: DOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: Myung In Pharm (Unknown)
Responsible Party: Principal Investigator, Yongcheol Kim, Clinical Associate Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9-2022-0141
Record Dates: First submitted 2023-01-06; First posted 2023-01-27 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Radiation Exposure
Keywords: DOSE
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Conventional Right Radial Artery Approach and Left Distal Radial Artery Approach for Coronary Angiography and Interventions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left distal radial artery approach (Experimental): Coronary angiography and intervention were performed using the left distal radial artery approach
  Interventions: Procedure: Radial Artery Puncture Method for Coronary Angiography and Intervention
- Right Radial Artery Approach (Active Comparator): Coronary angiography and intervention were performed using the Right Radial Artery Approach
  Interventions: Procedure: Radial Artery Puncture Method for Coronary Angiography and Intervention

INTERVENTIONS:
Procedure: Radial Artery Puncture Method for Coronary Angiography and Intervention — Radial Artery Puncture Method for Coronary Angiography and Intervention

SUMMARY:
The purpose of this study is to show that the radiation exposure of the left distal radial artery approach is superior to the conventional right radial artery approach in terms of less radiation exposure.

DETAILED DESCRIPTION:
The conventional radial approach is now recognized as the basic technique in coronary artery surgery. Compared to the femoral artery access, the main advantage is the increased stability due to the reduction of massive bleeding. Due to these advantages, recent guidelines recommend the conventional radial approach as the basic approach for all acute myocardial infarction (AMI) cases with or without ST-segment elevation. In particular, in the case of ST-segment elevation myocardial infarction (STEMI), new antiplatelet agents such as Ticagrelor and Prasugrel and strong antiplatelet agents such as Glycoprotein inhibitors have been used to prevent major vascular complications. For these many operators, primary percutaneous coronary intervention (PCI) through the radial artery is recommended. At this time, the operator prefers the right radial artery approach because of the comfort of performing the procedure on the patient's right side. However, the operator sometimes has to substitute the left radial artery or femoral artery access due to difficulty in manipulating the catheter due to severe tortuousness of the right subclavian artery. Although the left radial artery approach requires less operation time and radiographic imaging time due to less tortuousness of the left subclavian artery, the right conventional radial approach is still preferred due to the ergonomic inconvenience of having to lean toward the patient. Patients undergoing coronary angiography (CAG) were randomly assigned to the left snuffbox approach and the right conventional radial approach, and the surgeons' radiation exposure between the two approaches was evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 20 years or older
2. Patients scheduled for coronary angiography and intervention

Exclusion Criteria:

1. When the pulse of the Left distal radial artery cannot be palpated
2. When the pulse of the right conventional radial artery cannot be palpated
3. In case of arteriovenous fistula
4. Acute myocardial infarction (AMI) patients
5. In case femoral artery access must be performed (state of shock, etc.)
6. In case of atrioventricular block
7. When an ergonovine provocation test is required
8. When the patient refuses to consent to the study
9. a pregnant or nursing woman

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Radiation exposure examination | Through procedure completion, up to 24 hours
  Radiation exposure for surgeons in the case of the left distal radial artery approach and the right radial artery approach, respectively

SECONDARY OUTCOMES:
Fluoroscopy time | Through procedure completion, up to 24 hours
  Fluoroscopy time
Corrected by X-ray dose Radiation exposure of surgeons | Through procedure completion, up to 24 hours
  Corrected by X-ray dose Radiation exposure of surgeons
Corrected by X-ray dose Radiation | Through procedure completion, up to 24 hours
  Corrected by X-ray dose Radiation
Hemostasis time | Through procedure completion, up to 24 hours
  Hemostasis time
Procedure success rate | Through procedure completion, up to 24 hours
  Procedure success rate
Amount of contrast agent used | Through procedure completion, up to 24 hours
  Amount of contrast agent used

CONTACTS AND LOCATIONS:
Overall Officials: Yongcheol Kim, MD, PhD, Study Director — Severance Hospital
Locations (3):
- South Korea (3):
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong, Gyeonggi-do
  - Yongin Severance Hospital, Yongin, Gyeonggi-do

IPD SHARING:
Plan to Share IPD: No